CLINICAL TRIAL: NCT07261267
Title: The Effect of Music Therapy on the Radiotherapy Experience of Cancer Patients Undergoing Radiotherapy: A Randomised Controlled Trial
Brief Title: Music Therapy's Effect on Cancer Patients Undergoing Radiotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Ünal Önsüz, Lecturer, PhD, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17.07.2025 - 2025/1
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Radiotherapy
Keywords: Music Therapy; Radiotherapy; Anxiety; Pain; Stress
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Pain | interventions — Music Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy Group (Experimental Arm) (Experimental): Description: Consists of patients receiving curative radiotherapy (RT) who receive the music therapy intervention in addition to standard care to improve their radiotherapy experience.
  Interventions: Other: Music Therapy
- Control Group (Standard Care Arm) (Active Comparator): Description: Consists of patients receiving curative radiotherapy (RT) who receive only the standard radiation oncology care as per hospital protocol during their treatment.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Other: Music Therapy — Intervention: A personalized 15-20 minute music listening session is administered by a certified music therapist during the first session of radiotherapy.
  Patients select from a list of meditative, instrumental (wordless), and music that lacks peaks (sudden attacks).
  Music is presented via headphones before the session and as ambient listening during the session.
  Arms: Music Therapy Group (Experimental Arm)
Other: Standard Care (in control arm) — Intervention: These patients do not receive the music therapy intervention during their radiotherapy treatment.
  Arms: Control Group (Standard Care Arm)

SUMMARY:
The goal of this randomized controlled clinical study is to learn about the effects of music therapy on anxiety, stress, pain, and patient satisfaction in cancer patients who are newly starting radiotherapy (radiation treatment).

The main questions it aims to answer are:

Can music therapy lower the levels of anxiety and stress in patients receiving radiotherapy? Can music therapy improve the pain felt during the radiotherapy experience and overall satisfaction? Researchers will compare patients receiving standard radiotherapy (control group) with patients receiving music therapy alongside their radiotherapy (experimental group).

Participants (72 total) will:

Be 18 years and older and newly starting curative radiotherapy. Answer short surveys (STAI-SF, SDT, VAS) to measure their anxiety, stress, and pain levels before and after treatment.

Participants in the experimental group will receive a 15-20 minute music therapy session consisting of meditative and instrumental music during their first radiotherapy session.

This study aims to provide reliable data to guide clinical practice by showing whether music therapy offers a multifaceted approach to managing the psychological and physical challenges associated with cancer treatment.

DETAILED DESCRIPTION:
This study is a single-blind randomized controlled trial 20202020evaluating the effect of music therapy in managing the emotional and physical difficulties experienced by cancer patients who are newly starting curative radiotherapy (RT).Study Site: The study will take place at the Kocaeli University Hospital Radiation Oncology Unit.Objectives: The primary aim is to examine the effect of music therapy on anxiety, stress, pain, and patient satisfaction, and to determine how it can improve the RT experience.Intervention Application:Timing and Duration: Music therapy will be administered during the first RT session in sessions lasting 15-20 minutes. (Literature reports that $<20$ minutes reduces anxiety ).Provider: The intervention will be administered by a certified music therapist. Music Selection: Patients will be asked to choose music that has a meditative effect, is instrumental (without lyrics), and lacks peaks (sudden attacks), based on their preference and inclination. The music options provided will include Far Eastern music, music accompanied by a light-beat rhythm instrument (bendir), Ney-heavy Mesnevi music with meditative effects, and meditative Saba makam music.Listening Method: The patient's selected music will be played via headphones for 15 minutes before the session, and as ambient listening during the session. For patients with head and neck or brain cancer, only ambient listening will be used during the procedure for consistency.Data Collection and Timeline:Measurement Location: Measurements will be taken by researchers at the Kocaeli University Radiation Oncology Unit.Study Duration: The study starts on December 1, 2025, and ends on January31, 2026, with a total duration of 7 months.

Statistical Analysis:The collected data will be analyzed using the following methods: Between-group comparisons: Independent Sample T-test or Mann-Whitney U test37.Pre-post changes: Repeated Measures ANOVA.The significance level is set at $p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Must be a cancer patient 18 years of age or older.
* Must be newly starting curative external radiotherapy.
* Must volunteer to participate in the study and sign the Informed Consent form.

Exclusion Criteria:

* Having an advanced stage psychiatric disorder (e.g., schizophrenia).
* Having hearing loss.
* Having a prior history of an adverse reaction to music therapy.
* Receiving radiotherapy for palliative (symptom relief) purposes.
* Having received radiotherapy previously (for reasons such as brachytherapy, a different type of cancer, or recurrence).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety Level (STAI-SF) | mmediately before the start of the radiotherapy session (Pre-test) and immediately after the end of the radiotherapy session (Post-test).
  ssessment of the effect of the music therapy intervention on the anxiety levels of cancer patients receiving curative radiotherapy, using the State-Trait Anxiety Inventory-Short Form (STAI-SF). The measured difference will be compared between the intervention group and the control group.
Change in Stress Level (SDT) | Immediately before the start of the radiotherapy session (Pre-test) and immediately after the end of the radiotherapy session (Post-test).
  Assessment of the effect of the music therapy intervention on the general distress/stress levels experienced by cancer patients receiving curative radiotherapy, using the Symptom Distress Thermometer (SDT). The measured difference will be compared between the intervention group and the control group.

SECONDARY OUTCOMES:
Change in Procedural Pain Level (VAS) | Immediately before the start of the radiotherapy session (Pre-test) and immediately after the end of the radiotherapy session
  Assessment of the effect of the music therapy intervention on the severity of pain felt during or related to the radiotherapy procedure, using the Visual Analog Scale (VAS). The measured difference will be compared between the groups.
Patient Satisfaction Level (VAS) | Immediately after the end of the radiotherapy session (Post-test).
  Assessment of the effect of the music therapy intervention on patients' overall satisfaction levels with their radiotherapy experience, using the Visual Analog Scale (VAS). Satisfaction scores will be compared between the groups.

OTHER OUTCOMES:
Baseline Information Level (EORTC QLQ-INFO25) | At the start of the study (Pre-test).
  Determination of the baseline Information Levels of enrolled patients using the EORTC QLQ-INFO25. This is used to assess baseline similarity between groups, and the potential effect of the information level on other parameters will also be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The specific IPD to be shared includes all individual, anonymized patient data collected in the study. This data comprises:
  Demographic Data (such as age and gender).
  Disease and Treatment Information (such as cancer type, RT start date).
  Data from All Scales Used (STAI-SF, SDT, VAS Pain, VAS Satisfaction, and EORTC QLQ-INFO25 scores).
  The data will be coded to exclude any direct identifiers that could reveal the participants' identity.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Yang HF, Chang WW, Chou YH, Huang JY, Liao YS, Liao TE, Tseng HC, Chang ST, Chen HL, Ke YF, Tsai PF, Chan HM, Chang BJ, Hwang YT, Tsai HY, Lee YC. Impact of background music listening on anxiety in cancer patients undergoing initial radiation therapy: a randomized clinical trial. Radiat Oncol. 2024 Jun 11;19(1):73. doi: 10.1186/s13014-024-02460-3. PMID 38862982
- [Background] Wilson JM, Franqueiro AR, Edwards RR, Chai PR, Schreiber KL. Individuals with fibromyalgia report greater pain sensitivity than healthy adults while listening to their favorite music: the contribution of negative affect. Pain Med. 2024 May 2;25(5):352-361. doi: 10.1093/pm/pnae005. PMID 38291916
- [Background] Terzi, E. (2022). The effect of listening to music with or without patient selection on pain during cesarean section and its contribution to anesthesia technicians. Journal of Experimental and Clinical Medicine, 39(3), 786-792.
- [Background] Tao WW, Jiang H, Tao XM, Jiang P, Sha LY, Sun XC. Effects of Acupuncture, Tuina, Tai Chi, Qigong, and Traditional Chinese Medicine Five-Element Music Therapy on Symptom Management and Quality of Life for Cancer Patients: A Meta-Analysis. J Pain Symptom Manage. 2016 Apr;51(4):728-747. doi: 10.1016/j.jpainsymman.2015.11.027. Epub 2016 Feb 12. PMID 26880252
- [Background] Gulbahar Ates S, Demirel BB, Kekilli E, Ozturk E, Ucmak G. Primary tumor heterogeneity on pre-treatment [68Ga]Ga-PSMA PET/CT for the prediction of biochemical recurrence in prostate cancer. Rev Esp Med Nucl Imagen Mol (Engl Ed). 2024 Nov-Dec;43(6):500032. doi: 10.1016/j.remnie.2024.500032. Epub 2024 Aug 2. PMID 39097169
- [Background] Hewis J. Music and Music Therapy in the Medical Radiation Sciences. J Med Imaging Radiat Sci. 2018 Dec;49(4):360-364. doi: 10.1016/j.jmir.2018.09.009. Epub 2018 Oct 23. No abstract available. PMID 30514551
- [Background] Jiang X, Gao J, Zheng Y. Effectiveness of traditional Chinese medicine music therapy on anxiety and depression emotions of lung cancer patients: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2021 Mar 26;100(12):e25040. doi: 10.1097/MD.0000000000025040. PMID 33761662
- [Background] Imani M, Jalali A, Salari N, Abbasi P. Effect of instrumental music on anxiety and depression among hemodialysis patients: A randomized controlled trial. J Educ Health Promot. 2021 Aug 31;10:305. doi: 10.4103/jehp.jehp_1472_20. eCollection 2021. PMID 34667805
- [Background] Forbes E, Baker AL, Britton B, Clover K, Skelton E, Moore L, Handley T, Oultram S, Oldmeadow C, Gibberd A, McCarter K. A systematic review of nonpharmacological interventions to reduce procedural anxiety among patients undergoing radiation therapy for cancer. Cancer Med. 2023 Oct;12(20):20396-20422. doi: 10.1002/cam4.6573. Epub 2023 Oct 6. PMID 37803922
- [Background] Fernando GVMC, Wanigabadu LU, Vidanagama B, Samaranayaka TSP, Jeewandara JMKC. "Adjunctive Effects of a Short Session of Music on Pain, Low-mood and Anxiety Modulation among Cancer Patients" - A Randomized Crossover Clinical Trial. Indian J Palliat Care. 2019 Jul-Sep;25(3):367-373. doi: 10.4103/IJPC.IJPC_22_19. PMID 31413450
- [Background] Chen HH, Lai CH, Hou YJ, Kuo LT. The Efficacy of Music Intervention in Patients with Cancer Receiving Radiation Therapy: A Systematic Review and Meta-Analysis. Cancers (Basel). 2025 Feb 18;17(4):691. doi: 10.3390/cancers17040691. PMID 40002284